CLINICAL TRIAL: NCT03384849
Title: Clinical Evaluation of a Fiber-optic Sensor System for Monitoring Respiration Activity and Heart Work During MRI Examinations
Brief Title: Evaluation of an MRI-compatible Vital Signs Sensor System
Acronym: OPTO-MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Military Institute of Aviation Medicine (Other Government)
Responsible Party: Sponsor
Other Study IDs: OPTO-MRI_01/2017
Record Dates: First submitted 2017-12-20; First posted 2017-12-27 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Anxiety; Claustrophobia; Hyperventilation; Stress
Keywords: Fiber-optic sensor system; Magnetic resonance imaging; Medical monitoring; Physiological parameters
MeSH Terms: conditions — Anxiety Disorders; Claustrophobia; Hyperventilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRI patients: Up to 200 patients of different age, weight and sex, which undergo MRI examinations.
  Interventions: Diagnostic Test: MRI examination

INTERVENTIONS:
Diagnostic Test: MRI examination — The part of the body that is being scanned and the time of the MRI examination are not relevant.

SUMMARY:
This study is to determine the possibility of assessing the level of anxiety in MRI patients by means of the respiration rate (RR) and heart rate (HR) indicators acquired by a fiber-optic sensor system. The mean RR and/or HR values recorded at the beginning and the end of an MRI scanning will be referred to the State Trait Anxiety Inventory (STAI) scores completed before and after the MRI scanning, respectively.

DETAILED DESCRIPTION:
The main purpose of the study is to determine the possibility of assessing the level of anxiety by means of the respiration curve and/or ballistocardiographic (BCG) signal acquired from MRI patients using a fiber-optic sensor system. In many patients, the MRI examination causes enormous stress due to limited space in the scanner, isolation during the examination and high noise levels. Usually, anxiety or stress triggers an increase in respiration rate (RR), leading to hyperventilation in extreme cases. There are also frequent cases of disturbances in heart rate (HR). Thus, the symptoms of claustrophobia can be detected by monitoring respiration activity and heart work.

The fiber-optic sensor system consists of a sensor mat, an interrogator and a personal computer (PC), and records respiratory and BCG signals in patients during MRI. The metal-free sensor mat is placed under the patient's back, does not pose a threat to the patient and has no influence over the quality of imaging. The interrogation module detects the optical signal including vital signs, and the PC with software developed for signal processing and visualization enable the MRI operator to monitor patient's RR and HR.

Up to 200 MRI patients in different age, weight, and gender will be participated in the study. They will be asked to complete the State Trait Anxiety Inventory (STAI) questionnaire in order to estimate anxiety level before and after the MRI scanning. Relations between the STAI X-1 scores and the mean RR and/or HR values recorded at the beginning and the end of the MRI scanning will be analyzed using descriptive statistic methods. The research scheme includes also the collection of the STAI X-2 scores before the MRI scanning. Finally, the values of the physiological parameters, which may indicate a dangerous level of anxiety will be determined. Positive results of the clinical evaluation will predestine the fiber-optic sensor system to be implemented in routine MRI procedures.

ELIGIBILITY:
Inclusion Criteria:

* MRI patients

Exclusion Criteria:

* Same as in MRI procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 200 MRI patients of different age, weight and sex.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01-03 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Optical signal | 60 minutes
  Instantaneous spectral position of the fiber Bragg grating (FBG) reflection peak in nanometers that represents respiration curve and ballistocardiogram

SECONDARY OUTCOMES:
RR | 60 minutes
  Respiration rate in respirations per minute
HR | 60 minutes
  Heart rate in beats per minute

OTHER OUTCOMES:
RR_1 | 2 minutes
  Respiration rate at the beginning of the MRI scanning in respirations per minute
RR_2 | 2 minutes
  Respiration rate at the end of the MRI scanning in respirations per minute
HR_1 | 2 minutes
  Heart rate at the beginning of the MRI scanning in beats per minute
HR_2 | 2 minutes
  Heart rate at the end of the MRI scanning in beats per minute
STAI X-1_1 | 1 minute
  STAI X-1 scores completed before the MRI scanning. Scale range: 20 - 80 (raw scores), where 20 means low anxiety, and 80 indicates high anxiety (the higher the result, the higher the level of anxiety).
STAI X-1_2 | 1 minute
  STAI X-1 scores completed after the MRI scanning. Scale range: 20 - 80 (raw scores), where 20 means low anxiety, and 80 indicates high anxiety (the higher the result, the higher the level of anxiety).
STAI X-2 | 1 minute
  STAI X-2 scores completed before the MRI scanning. Scale range: 20 - 80 (raw scores), where 20 means low anxiety, and 80 indicates high anxiety (the higher the result, the higher the level of anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Dziuda, DSc, PhD, Principal Investigator — Military Institute of Aviation Medicine
Locations (1):
- Military Institute of Aviation Medicine, Warsaw, Poland

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-01-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT03384849/Prot_SAP_ICF_000.pdf